CLINICAL TRIAL: NCT02505854
Title: Influence of Probiotic and Symbiotic in Body Weight, Blood Sugar and Lipemia of Obese Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal do Rio de Janeiro (Other)
Collaborators: Rio de Janeiro State Research Supporting Foundation (FAPERJ) (Other Government)
Responsible Party: Principal Investigator, Louise Crovesy de Oliveira, Principal investigator, Universidade Federal do Rio de Janeiro
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CEP 104-14
Record Dates: First submitted 2015-07-16; First posted 2015-07-22 (Estimated); Last update posted 2019-12-10 (Actual); Status verified 2019-12

CONDITIONS: Obesity
Keywords: Obesity; Probiotic; Symbiotic; Weight loss; Gut microbiota; Bifidobacterium lactis; Fructooligosaccharide; Blood sugar; Lipemia; Metabolome
MeSH Terms: conditions — Obesity; Weight Loss; Hyperlipidemias | interventions — Probiotics; fructooligosaccharide; Gelatin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Probiotic (Active Comparator): Hypocaloric diet associated with capsule containing 1billion UFC Bifidobacterium lactis and sache with 5 g of maltodextrin
  Interventions: Dietary Supplement: Probiotic
- Symbiotic (Active Comparator): Hypocaloric diet associated with capsule containing 1billion UFC Bifidobacterium lactis and sache with 5 g of fructooligosaccharide
  Interventions: Dietary Supplement: Symbiotic
- Placebo (Placebo Comparator): Hypocaloric diet associated with capsule containing 50g of gelatin and sache with 5 g of maltodextrin
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotic — Hypocaloric diet associated with capsule containing 1billion UFC Bifidobacterium lactis and sache of maltodextrin
  Other Names: Bifidobacterium lactis
  Arms: Probiotic
Dietary Supplement: Symbiotic — Hypocaloric diet associated with capsule containing 1billion UFC Bifidobacterium lactis and sache of fructooligosaccharide
  Other Names: Bifidobacterium lactis and fructooligosaccharide
  Arms: Symbiotic
Dietary Supplement: Placebo — Hypocaloric diet associated with capsule containing 50g of gelatin and sache of maltodextrin
  Other Names: Gelatin
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate whether gut microbiota modulation by probiotic and symbiotic contribute with weight loss and improvement of metabolic parameters in women with obesity.

DETAILED DESCRIPTION:
We will evaluate the effects of probiotic and symbiotic on weigh loss, blood glucose, lipid profile, metabolomic profile, and gut microbiota composition variables in women with obesity.

ELIGIBILITY:
Inclusion Criteria:

* Women;
* Adult;
* Obese (BMI between 30 and 39,9 Kg/m²).

Exclusion Criteria:

* Pregnancy or nursing;
* Smokers;
* Drinkers;
* Use of drug or phytotherapic;
* Diagnosis of any cronic disease;
* Daily consumption of yogurt.

Ages: 25 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2018-11 (Actual)

PRIMARY OUTCOMES:
Evaluate the effect of probiotic and symbiotic on weight loss of women obese | Baseline and 60 days and 15 days after the end of the intervention
  Determine and evaluate change in body weight and body mass index after intervention.

SECONDARY OUTCOMES:
Effect of probiotic and symbiotic on blood glucose | Baseline, 60 days and 15 days after the end of the intervention
  Determine and comparing the blood glucose in plasma before and after intervention
Effect of probiotic and symbiotic on insulin resistance | Baseline and 60 days
  Compare insulin resistance through HOMA-IR calculation before and after intervention and evaluate whether the intervention improvement in this parameter.
Effect of probiotic and symbiotic on lipid profile | Baseline and 60 days
  Compare lipid profile (total cholesterol, low-density lipoprotein, high-density lipoprotein, very low-density lipoprotein, triglyceride) in serum of blood before and after intervention and evaluate whether the intervention improvement in this parameter.
Effect probiotic and symbiotic on blood pressure | Baseline,60 days and 15 days after intervention conclusion
  Determine blood pressure and evaluate whether the intervention improvement blood pressure.
Effect of probiotic and symbiotic on gut microbiota composition | Baseline, 60 days and 15 days after intervention conclusion
  Determine and comparing the amount filos (Fimicutes, Bacteroidetes, Actinobacteria, Verrucomicrobia e Proteobacteria) in gut microbiota and whether the change in microbiota composition continue after stop probiotic and symbiotic intake
Effect of probiotic and symbiotic on stool consitency by Bristol scale | Baseline,60 days and 15 days after intervention conclusion
  Determine and comparing the stool consistency by Bristol scale. The Bristol scale is composed of 7 different stool consistency, being 1 and 2 lumpy, 3 and 4 normal, 5 to 7 loose.
Effect of probiotic and symbiotic on gastrointestinal symptons | Baseline,60 days and 15 days after intervention conclusion
  Evaluate the presence of gastrointestinal symptoms related to the probiotic and symbiotic. The gastrointestinal symptoms analyzed were abdominal pains, abdominal distension and abdominal discomfort, flatus, borborygmus using the Likert scale of 5 point, which 0 is absence of symptom and 4 is every day.
Effect of probiotic and symbiotic on metabolomic profile | Baseline and 60 days
  Determine and comparing change in metabolomic profile before and after intervention. The metabolomic profile was evaluated in the serum of blood Bruker DRX 500 MHz equipment (Bruker Spectrospin, Karlsruhe, Germany) generating hydrogen isotope 1 (1H)-NMR spectra, that was compared to database Human Metabolome Data Base.

CONTACTS AND LOCATIONS:
Overall Officials: Louise C Oliveira, MD student, Principal Investigator — Universidade Federal do Rio de Janeiro
Locations (1):
- Louise Crovesy de Oliveira, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Crovesy L, El-Bacha T, Rosado EL. Modulation of the gut microbiota by probiotics and symbiotics is associated with changes in serum metabolite profile related to a decrease in inflammation and overall benefits to metabolic health: a double-blind randomized controlled clinical trial in women with obesity. Food Funct. 2021 Mar 15;12(5):2161-2170. doi: 10.1039/d0fo02748k. PMID 33565558
- See also: Institute of Nutrition Josué de Castro — http://www.nutricao.ufrj.br/